CLINICAL TRIAL: NCT03915483
Title: Cognitive Transfer Effects on Working Memory and Higher Cognitive Functions by Combined Attentional Filter Exercise and tDCS in Healthy Younger Adults
Brief Title: Transfer Effects of Combined Attentional Filter Exercise and Transcranial Direct Current Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: German Center for Neurodegenerative Diseases (DZNE) (Other)
Responsible Party: Principal Investigator, Notger Müller, Prof. Dr. med. (Head of Neuroprotection Lab at the DZNE), German Center for Neurodegenerative Diseases (DZNE)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD021.1
Record Dates: First submitted 2019-04-08; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Healthy
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS group (Experimental): one session of computerized change detection attentional filter exercise (selective attention) combined with real tDCS
  Interventions: Device: transcranial direct current stimulation (tDCS)
- sham group (Sham Comparator): one session of computerized change detection attentional filter exercise (selective attention) combined with sham tDCS
  Interventions: Device: transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — sham or real tDCS for 10 minutes of 1.5 milliampere (mA) tDCS targeting the prefrontal and the posterior parietal cortex

SUMMARY:
Investigation of how a single session of an attentional filter exercise of distractor inhibition combined with tDCS modulates cognitive functions like working memory, decision making and attentional control.

DETAILED DESCRIPTION:
The study is designed as a between subject design with two groups defined by real or sham tDCS. The distractor inhibition exercise is conducted under either sham or real tDCS. Cognitive performance is assessed pre and post tDCS application, complemented by a short-termed follow-up on a consecutive day. Interindividual working memory capacity at baseline is taken into consideration.

ELIGIBILITY:
Inclusion Criteria:

* right-handed
* aged between 18 and 30 years
* normal or corrected to normal vision
* German-speaking

Exclusion Criteria:

* dyschromatopsia
* neurological or neuropsychiatric diseases
* low seizure threshold
* neurological medication
* metal implants in the head

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Performance change in computerized attentional filter exercise | 45 minutes on 1st day (pre) and on consecutive day (post)
  attentional filtering performance (in % correct), effects of distractor interference for different set sizes
Reaction change in computerized attentional filter exercise | 45 minutes on 1st day (pre) and on consecutive day (post)
  reaction times (in milliseconds), effects of distractor interference for different set sizes
Performance change in working memory and filtering performance | 30 minutes per pre-assessment, post assessment directly after intervention and short-termed follow-up on the consecutive day
  Working memory and filtering performance (in % correct), effects of distractor interference for different set sizes
Reaction change in working memory and filtering performance | 30 minutes per pre-assessment, post assessment directly after intervention and short-termed follow-up on the consecutive day
  reaction times (in milliseconds), effects of distractor interference for different set sizes

SECONDARY OUTCOMES:
Spatial Span | 10 minutes per pre-assessment and short-termed follow-up on the consecutive day
  computerized spatial span forward and backward
Iowa Gambling Task | 7 minutes per pre-assessment, post assessment directly after intervention and short-termed follow-up on the consecutive day
  Decision making performance
Trait-Anxiety | 2 minutes on first day
  Assessment of trait anxiety via State-Trait-Anxiety-Inventory on first day
State-Anxiety | 2 minutes on first and consecutive day
  Daily assessment of state anxiety via State-Trait-Anxiety-Inventory at the beginning of each testing day
Assessment of Sleep Quality | 10 minutes on first and consecutive day
  daily questionnaire assessing subjective rating of sleep of the previous night on 5- to 7-point Likert format and open questions (subjective quality of sleep, current fatigue, duration of sleep); no total score
Daily Performance Questionnaires | 5 minutes on first and consecutive day
  self developed questionnaire assessing subjective performance in tested paradigms (5-point Likert format); no total or sub score; Question 1: How difficult would you rate the task? (lowest (1) = very difficult; highest (5) = very easy) Question 2: Do you think your performance changed in the course of the task? (lowest (1) = strongly worsened; highest (5) = strongly improved)
Daily Strategy Questionnaires | 5 minutes on first and consecutive day
  reporting of used strategies in tested paradigms (open questions; subjects reported in written notes); self developed questionnaire for qualitative analyses of task demands; no scores; Question: Did you use a strategy? If so, please explain shortly.

CONTACTS AND LOCATIONS:
Overall Officials: Notger Müller, Prof. Dr., Principal Investigator — German Center for Neurodegenerative Diseases (DZNE)
Locations (1):
- German Center for Neurodegenerative Diseases, Magdeburg, Saxony-Anhalt, Germany

IPD SHARING:
Plan to Share IPD: No